CLINICAL TRIAL: NCT06416943
Title: Effects of a 3D-Printed Port-A Catheter Model Training Course for New Staff
Brief Title: 3D Port-A Catheter Model for New Staff
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fu Jen Catholic University (Other)
Responsible Party: Principal Investigator, Ke-Yun, Chao, Group leader of Respiratory Therapists, Fu Jen Catholic University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FJUH112278-2
Record Dates: First submitted 2024-05-12; First posted 2024-05-16 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Personal Satisfaction; Cancer
Keywords: 3D printed model; port-a catheter; nursing skill education
MeSH Terms: conditions — Personal Satisfaction; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3D medical education model group (Experimental): Received a regular learning plus 3D printing model
  Interventions: Other: 3D printed educational model

INTERVENTIONS:
Other: 3D printed educational model — Slide-based presention plus 3D printed port-A catheter model

SUMMARY:
The aim of this study is to develop a highly realistic 3D-printed Port-A catheter upper body model to enhance the effectiveness of training new nursing staff in Port-A catheter placement and care skills.

DETAILED DESCRIPTION:
Background： Cancer patients often require long-term administration of chemotherapy drugs, nutritional supplementation, and blood transfusions. During these treatments, an implantable central venous access (port-a catheter) is often utilized to avoid the inconvenience of repeated needle insertions for treatment and to minimize the risk of medication leakage. Port-A catheters are considered a safer clinical measure. However, poor care and maintenance of the catheter can lead to complications such as infection, catheter damage, and leakage, which can even result in death. Proper care and maintenance are crucial for the successful use of Port-A catheters. For nursing staff, acquiring professional knowledge in Port-A catheter care is essential for improving the quality of cancer patient care. Insufficient education and training in Port-A catheter care can lead to clinical errors that endanger patients' lives.

Methods： This study involves providing training to participants and assessing their performance and effectiveness. It employs a prospective quasi-experimental design with a single group and pre- and post-test evaluations. The study includes 50 newly recruited nursing staff.

Effect： The investigators anticipate that the use of a 3D-printed upper body Port-A catheter model will yield better results in the training of newly recruited nursing staff.

ELIGIBILITY:
Inclusion Criteria:

* New nursing staff joined Fu Jen Catholic University Hospital.

Exclusion Criteria:

* Refused to participate in the study.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Examination score of pre-intervention | pre-intervention
  score of pre-intervention (maximun 100 and minimum 0), higher means a better outcome.
Examination score of post-intervention | immediately after the intervention
  score of post-intervention (maximun 100 and minimum 0), higher means a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ke-Yun Chao, PhD, Principal Investigator — Fu Jen Catholic University Hospital
Locations (1):
- Fu Jen Catholic University Hospital, Fu Jen Catholic University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No